CLINICAL TRIAL: NCT03209570
Title: A Pilot Clinical Trial of TENA Identifi in the Nursing Home Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insight Therapeutics, LLC (Other)
Collaborators: Essity Hygiene and Health AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INSI-201706
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence, nursing home
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TENA Identifi with sensor wear data (Experimental): All individuals in this arm will receive care planning using TENA Identifi sensor wear data
  Interventions: Other: Care planning using TENA Identifi sensor wear data
- TENA Identifi without sensor wear data (Active Comparator): All individuals in this arm will receive care planning without using TENA Identifi sensor wear data
  Interventions: Other: Care planning without using TENA Identifi sensor wear data

INTERVENTIONS:
Other: Care planning using TENA Identifi sensor wear data — All individuals in this arm will receive TENA Identifi sensor wear and will have data available for care planning.
  Arms: TENA Identifi with sensor wear data
Other: Care planning without using TENA Identifi sensor wear data — All individuals in this arm will receive TENA Identifi sensor wear but the sensor wear data will not be used for care planning.
  Arms: TENA Identifi without sensor wear data

SUMMARY:
The purpose of this study is to prospectively compare a standard of care manual toileting protocol (e.g., "check and change" strategy) to toileting patterns recorded by the TENA Identifi system in identifying incontinence patterns and events, and, whether such data differentially improve a care planning strategy, nursing effort, product use, and wet-time for urinary incontinence.

DETAILED DESCRIPTION:
Urinary incontinence in nursing homes influences resident dignity and quality of life. It also drives significant use of healthcare resources, including time and caregiver assistance, and costs of care. Various toileting programs are used to address urinary incontinence, including habit training, bladder training, prompted voiding, and check and change procedures. Clinical trials have found that 33% to 60% of residents either became continent or reduced the frequency of incontinence episodes to less than one per day with the introduction of a prompted voiding program.

There are several drawbacks to current programs. Manually recorded wet checks do not identify when incontinence occurs, only when wetness is detected, reducing the precision of time of incontinence to the window of time between checks. Nursing home staff create individualized care plans for each resident, based on standard check and change procedures, but poor precision in ascertaining timing and quantity of incontinence episodes can contribute to less frequent resident toileting or changing.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 55 years of age or older with stable clinical status
2. Long-stay status (more than 90 days)
3. Ambulatory and able to use a toilet either independently or with assistance
4. Minimum Data Set (MDS) Level 1 (occasionally), 2 (frequently) or 3 (always) rating of incontinence
5. Currently wearing disposable briefs for urinary incontinence

Exclusion Criteria:

1. Chronically bed-bound (MDS G0110A rating 8)
2. MDS self-performance rating of 4 (total dependence) for toilet use
3. Fecal incontinence (MDS H0400 rating 0)
4. Use of urinary appliance such as catheters or ostomies (MDS H0100 Z)
5. Private duty nurse care
6. Residents who tear at clothing or disposable undergarments
7. Current urinary tract infection receiving treatment
8. Current diarrhea receiving treatment
9. Residents who are not likely to benefit from a toileting plan based on assessment of nursing staff

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-08-11 (Actual); Study Completion 2018-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Gravenstein, MD, MPH, Principal Investigator — Brown University; H Edward Davidson, PharmD, MPH, Principal Investigator — Insight Therapeutics, LLC
Locations (5):
- United States (5):
  - Chesapeake Health & Rehabilitation Center, Chesapeake, Virginia
  - Norfolk Health & Rehabilitation Center, Norfolk, Virginia
  - Insight Therapeutics, LLC, Norfolk, Virginia
  - Westminster-Canterbury on Chesapeake Bay, Virginia Beach, Virginia
  - Beth Sholom Village, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ouslander JG, Schnelle JF, Uman G, Fingold S, Nigam JG, Tuico E, Bates-Jensen B. Predictors of successful prompted voiding among incontinent nursing home residents. JAMA. 1995 May 3;273(17):1366-70. PMID 7715062
- [Background] Omli R, Skotnes LH, Romild U, Bakke A, Mykletun A, Kuhry E. Pad per day usage, urinary incontinence and urinary tract infections in nursing home residents. Age Ageing. 2010 Sep;39(5):549-54. doi: 10.1093/ageing/afq082. Epub 2010 Jul 14. PMID 20631404

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TENA Identifi With Sensor Wear Data | TENA Identifi Without Sensor Wear Data
Started | 24 | 25
Completed | 14 | 12
Not Completed | 10 | 13
Not completed — Death | 1 | 0
Not completed — Incomplete Data | 8 | 10
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TENA Identifi With Sensor Wear Data | TENA Identifi Without Sensor Wear Data | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 84.7 (14.5) | 79.4 (11.8) | 82.3 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 26
Height [Mean (Standard Deviation); unit: inches] | 64.6 (5.2) | 63.8 (3.8) | 64.2 (4.5)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.2 (7.23) | 25.9 (6.6) | 27.1 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Wet Events Per 24 Hours
Description: Comparison of the number of wet events per 24 hours as recorded by TENA Identifi, intervention versus control
Time Frame: 6 days
Population: The study design is a two group, two time-point, four site, randomized, longitudinal clinical trial. Means were generated by averaging the 3 daily counts in each assessment period (pre-intervention and post-intervention) for each group (control versus intervention).
Measure: Least Squares Mean (Standard Error); unit: events per 24 hours
Arm/Group | TENA Identifi With Sensor Wear Data | TENA Identifi Without Sensor Wear Data
Number analyzed (Participants) | 14 | 12
events per 24 hours
  Days 1-3 | 8.11 (1.31) | 5.75 (1.39)
  Days 7-9 | 7.05 (1.31) | 5.45 (1.39)

2. Secondary Outcome: Time Wet Per 24 Hours
Description: Comparison of the amount of time wet per 24 hours as recorded by TENA Identifi, intervention versus control
Time Frame: 6 days
Measure: Least Squares Mean (Standard Error); unit: hours per 24 hours
Arm/Group | TENA Identifi With Sensor Wear Data | TENA Identifi Without Sensor Wear Data
Number analyzed (Participants) | 14 | 12
hours per 24 hours
  Days 1-3 | 10.69 (1.83) | 9.70 (2.01)
  Days 7-9 | 10.24 (1.83) | 8.94 (2.01)

3. Secondary Outcome: Number of Brief Changes Per 24 Hours
Description: The number of brief changes per 24 hours, intervention versus control
Time Frame: 6 days
Measure: Least Squares Mean (Standard Error); unit: events per 24 hours
Arm/Group | TENA Identifi With Sensor Wear Data | TENA Identifi Without Sensor Wear Data
Number analyzed (Participants) | 14 | 12
events per 24 hours
  Days 1-3 | 3.25 (0.26) | 2.54 (0.28)
  Days 7-9 | 3.08 (0.26) | 2.52 (0.28)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 6 days/ two 72hr time periods (randomization through study completion)
Description: no additional adverse events were reported by nursing facilities
Arm/Group | TENA Identifi With Sensor Wear Data | TENA Identifi Without Sensor Wear Data
All-Cause Mortality (participants affected / at risk) | 1/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/12
Other Adverse Events (participants affected / at risk) | 0/14 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TENA Identifi With Sensor Wear Data (N=14) | TENA Identifi Without Sensor Wear Data (N=12)
Acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Resident was consented and randomized but passed away before sensor wear was placed on resident. No assessments occurred.

LIMITATIONS AND CAVEATS:
small sample size, lack of time and resources for facilities to assist with study, and resident's removing sensor wear.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/70/NCT03209570/Prot_SAP_000.pdf